CLINICAL TRIAL: NCT06228729
Title: Evaluation of the Association Between Electroencephalographic Changes and Hormonal Response to Tracheal Intubation and Surgical Stimulation in Abdominal Surgery: a Prospective Observational Study
Brief Title: Association Between EEG Changes and Hormonal Response to Tracheal Intubation and Surgical Stimulation
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyun-Kyu Yoon, Clinical assistant professor, Seoul National University Hospital
Other Study IDs: 2311-093-1484
Record Dates: First submitted 2024-01-18; First posted 2024-01-29 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Abdominal Surgery; Endotracheal Intubation; Surgical Incision; Electroencephalogram
MeSH Terms: conditions — Surgical Wound | interventions — Intubation, Intratracheal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Endotracheal intubation — Inserting endotracheal tube into the trachea

SUMMARY:
This study aims to prospectively evaluate the relationship between changes in EEG and hormonal responses induced by endotracheal intubation and surgical incision following general anesthesia.

DETAILED DESCRIPTION:
This study aims to investigate the relationship between changes in EEG patterns and stress hormone levels in patients undergoing open abdominal surgery under general anesthesia when subjected to endotracheal intubation and surgical incision stimuli.

Hormone measurements (cortisol, ACTH) are taken at four time points: before endotracheal intubation (T1), one minute after intubation (T2), and one minute after surgical incision (T3). The investigators evaluate the correlation between hormone levels (cortisol, ACTH) and EEG band power changes (alpha, beta, delta) before and after endotracheal intubation and surgical incision.

ELIGIBILITY:
Inclusion Criteria:

* 1) Patients scheduled to undergo open abdominal surgery under general anesthesia with endotracheal intubation.
* 2) Patients requiring invasive blood pressure monitoring during surgery

Exclusion Criteria:

* 1) Patients transferred to the intensive care unit after surgery
* 2) Surgery duration of less than one hour
* 3) Patients with neurological underlying conditions
* 4) Patients on chronic use of psychotropic medications and opioid drugs
* 5) Emergency surgery

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing open abdominal surgery and endotracheal intubation under general anesthesia
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-10-28 (Actual); Study Completion 2025-11-21 (Actual)

PRIMARY OUTCOMES:
Association between band power changes in EEG and hormone respones caused by endotracheal intubation | from the start of anesthesia induction to one minute after endotracheal intubation

SECONDARY OUTCOMES:
Association between band power changes in EEG and hormone respones caused by surgical incision | from the start of anesthesia induction to one minute after surgical incision

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea